CLINICAL TRIAL: NCT02632435
Title: A Pragmatic Randomized Trial Standard of Care Vascular Access Strategies for (Neo)Adjuvant Trastuzumab-based Breast Cancer Treatment OTT 15-06 A Study From the REthinking Clinical Trials Program (REaCT-vascular Access Trastuzumab Study).
Brief Title: Randomized Trial Standard of Care Vascular Access Strategies for (Neo)Adjuvant Trastuzumab-based Breast Cancer Treatment.
Acronym: OTT 15-06
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Ottawa Hospital Research Institute (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: 15-089
Record Dates: First submitted 2015-12-08; First posted 2015-12-16 (Estimated); Last update posted 2019-09-06 (Actual); Status verified 2019-08

CONDITIONS: Breast Cancer; Cancer
Keywords: HER2 positive
MeSH Terms: conditions — Breast Neoplasms; Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Peripherally inserted central catheter (Other): PICC line will be inserted for the delivery and duration of chemotherapy.
  Interventions: Device: PICC
- portacath (Other): PORT will be inserted for the delivery and duration of chemotherapy and trastuzumab.
  Interventions: Device: PORT

INTERVENTIONS:
Device: PICC — Participants will be randomized to a PICC for vascular access during chemotherapy.
  Arms: Peripherally inserted central catheter
Device: PORT — Participants will be randomized to a PORT for vascular access during chemotherapy
  Arms: portacath

SUMMARY:
In the REaCT-Vascular Access Trastuzumab study (REaCT-VA), the investigator will use a novel method to allow comparisons of established standard of care vascular access strategies using the "integrated consent model" as part of a pragmatic clinical trial. The investigator wishes to address a non-pharmacologic issue regarding standard of care vascular access devices. Peripherally inserted central catheters (PICC lines) versus subcutaneously implanted devices (PORTs).

ELIGIBILITY:
Inclusion Criteria

* Histologically confirmed primary breast cancer
* Planned to start trastuzumab based neo/adjuvant therapy: FEC-DH or AC-DH, or; dose-dense AC-TH, or docetaxel/cyclophosphamide/trastuzumab or docetaxel/carboplatin/trastuzumab, or weekly paclitaxel with trastuzumab.
* ≥19 years of age
* Able to provide verbal consent

Exclusion Criteria

• Contraindication to central line placement.

Min Age: 19 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 56 (Actual)
Dates: Start 2016-04; Primary Completion 2019-05 (Actual); Study Completion 2019-05 (Actual)

PRIMARY OUTCOMES:
Accrual rates | one year
  Percentage of patients who receive (neo)adjuvant IV systemic therapy with trastuzumab compared to the number of participants who agree to randomization.
Patient compliance | One year
  Percentage of participants who are randomized who accept randomization will be calculated.

SECONDARY OUTCOMES:
Physician engagement | One year
  Percentage of medical oncologists who have agreed to participate in the trial compared to the percentage who approached patients regarding the trial.
Rates of events | One year
  Rates of documented thrombotic events, need for anticoagulation, line infections, phlebitis, and extravasations during systemic therapy.

CONTACTS AND LOCATIONS:
Overall Officials: Mark Clemons, MD, Principal Investigator — The Ottawa Hospital
Locations (1):
- The Ottawa Hospital Cancer Centre, Ottawa, Ontario, Canada

REFERENCES:
- [Derived] Clemons M, Stober C, Kehoe A, Bedard D, MacDonald F, Brunet MC, Saunders D, Vandermeer L, Mazzarello S, Awan A, Basulaiman B, Robinson A, Mallick R, Hutton B, Fergusson D. A randomized trial comparing vascular access strategies for patients receiving chemotherapy with trastuzumab for early-stage breast cancer. Support Care Cancer. 2020 Oct;28(10):4891-4899. doi: 10.1007/s00520-020-05326-y. Epub 2020 Jan 30. PMID 32002617